CLINICAL TRIAL: NCT05287711
Title: Adjunctive Motivational Alcohol Intervention to Prevent Intimate Partner Violence
Brief Title: Adjunctive Motivational Alcohol Intervention to Prevent IPV
Acronym: MET-SAH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NURA-007-20F
Record Dates: First submitted 2022-03-09; First posted 2022-03-18 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Alcohol Use and Intimate Partner Violence
Keywords: Intimate Partner Violence; Alcohol Use
MeSH Terms: conditions — Alcohol Drinking | interventions — Motivational Interviewing; Ethanol; Therapeutics

STUDY DESIGN:
Intervention Model Description: Participants will receive motivational enhancement therapy for alcohol use problems and this will be compared to an alcohol psychoeducational intervention.
Who Masked: Outcomes Assessor
Masking Description: Assessors will be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Motivational Enhancement Therapy (Experimental): Motivational enhancement therapy for alcohol use problems, which includes empathic support, feedback and advice, strategies for enhancing self-efficacy, techniques for eliciting self-motivational statements from the participant, strategies for addressing participant ambivalence about change and participant resistance to change, and methods for eliciting and affirming commitment to a specific change plan (active intervention).
  Interventions: Behavioral: Motivational Enhancement Therapy; Behavioral: Strength at Home
- Alcohol Education Control (Experimental): Psychoeducational intervention intended to: (1) dispel myths about the effects of alcohol, (2) provide information about the general risks of drinking and process of recovery from alcohol problems, (3) provide information about the specific risks related to family relationships and IPV, (4) offer self-help program information and related strategies to address drinking problems, (5) promote and encourage healthy decision-making, and (6) reinforce the benefits of abstinence or controlled drinking.
  Interventions: Behavioral: Alcohol Education Control; Behavioral: Strength at Home
- Telephone Monitoring (Other): Brief supportive telephone monitoring sessions that are commonly delivered while Veterans wait to begin their groups (treatment as usual).
  Interventions: Behavioral: Treatment as Usual; Behavioral: Strength at Home

INTERVENTIONS:
Behavioral: Motivational Enhancement Therapy — In Session 1, the therapist provides personalized feedback on a range of assessment variables, including alcohol consumption levels, negative consequences from alcohol use, and family risk of alcoholism. Sessions 2-4 are follow-through sessions in which the therapist attempts to help the Veteran participant establish or reaffirm a commitment to an action plan for addressing alcohol concerns.
  Other Names: MET
  Arms: Motivational Enhancement Therapy
Behavioral: Alcohol Education Control — Will consist of 4 weekly individual sessions, approximately 60 minutes each. AE therapists will explain that their job is to provide the Veteran participants with information and education about the effects of alcohol, and that it is up to the Veteran participant to use this information as he sees fit. In each session, the Veteran participant will watch an educational videotape in a comfortable consulting room and will be given an opportunity to discuss the videotape with the project therapist for approximately 10 minutes. Written educational materials will supplement the information provided in the videos, and the therapist will ask several structured questions to determine whether the Veteran participant understood the material presented in the video.
  Other Names: AE
  Arms: Alcohol Education Control
Behavioral: Treatment as Usual — Supportive telephone monitoring sessions that ensure equal spacing between assessments across conditions and equal number of therapist contacts.
  Other Names: TAU
  Arms: Telephone Monitoring
Behavioral: Strength at Home — IPV intervention which consists of 12 weekly, 2-hour cognitive-behavioral sessions offered in a closed group format and co-led by doctoral level male and female therapists. Strength at Home is based on a social information processing model of trauma and IPV and provides material covering psychoeducation regarding trauma and IPV, conflict and anger management skills, assertiveness training, and skills in stress management and communication.
  Other Names: SAH

SUMMARY:
This is a study to provide much-needed experimental data on the efficacy of a brief alcohol Motivational Enhancement Therapy (MET) pre-group intervention for Veterans receiving group treatment for IPV perpetration. The investigators will compare those assigned to receive this 2-session MET intervention to those receiving a 2-session Alcohol Education (AE) intervention or a 2-session standard treatment as usual (TAU) telephone monitoring intervention. The investigators will examine whether MET leads to greater reductions in alcohol use problems and IPV perpetration, and increased help-seeking behavior for alcohol use problems. Participants will be 300 Veterans drawn from the Strength at Home IPV intervention program across the entire Veterans Health Administration system.

DETAILED DESCRIPTION:
Veterans exposed to trauma are at elevated risk for perpetration of intimate partner violence (IPV) and for the development of alcohol-related problems. Despite commonly found associations between alcohol misuse and IPV, the investigators are aware of no prior research in Veterans examining the impact of adjunctive alcohol interventions for those receiving IPV intervention. The investigators propose to provide much-needed experimental data on the efficacy of a brief 2-session alcohol Motivational Enhancement Therapy (MET) pre-group intervention for Veterans receiving group treatment for IPV perpetration. More specifically, the investigators propose to examine whether those assigned to receive this 2-session MET intervention, relative to those receiving a 2-session Alcohol Education (AE) intervention or a 2-session standard treatment as usual (TAU) telephone monitoring intervention, evidence greater reductions in alcohol use problems and IPV perpetration, and increased help-seeking behavior for alcohol use problems. Participants will be 300 Veterans drawn from the Strength at Home IPV intervention program across the entire Veterans Health Administration system. Participants will be randomized to their pre-group conditions and then assigned to Strength at Home groups for IPV, and will receive referrals for substance use treatment in the VA system or the community. Participants with clinically relevant alcohol use problems, as determined by baseline screening measures, will complete assessments of alcohol use, readiness to change, IPV and help-seeking behavior at baseline, post IPV intervention group (3 months after completion of 2-session alcohol intervention), and four separate 3-month follow-ups after the post-treatment assessment. Differences between conditions on the major outcome variables involving alcohol use, IPV, help-seeking, and treatment engagement will be examined with random-effects regression models using an intent-to-treat approach. Study findings may assist in enhancing the efficacy of IPV interventions for the Veteran population to help ensure the safety and well-being of Veterans and their families.

ELIGIBILITY:
Inclusion Criteria:

All Veteran participants must meet the following eligibility criteria:

* participant is a Veteran
* minimum age 18
* participant is enrolled in the Strength at Home program following program intake
* participant displays evidence of alcohol-related problems during program intake, as indicated by any of the following:

  * a report of physical IPV while under the influence of alcohol in the past year
  * a score of 8 or greater on the Alcohol Use Disorders Identification Test (AUDIT)
  * consumption of 6 or more standard drinks per occasion on one or more occasions in the previous 6 months
  * average weekly consumption of 14 or more standard drinks in the prior 6 months
* participant provides written consent to participate in the study
* inclusion for this study is broad because this is a population who possesses a number of comorbid problems and exclusion for those based on psychopathology or risk for aggression could potentially lead to a biased sample

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Quantity/Frequency of Alcohol Consumption, Self-Report (QFV) | Baseline, post-treatment, three-month, six-month, nine-month, and twelve-month follow-ups
  Participants will be shown a standard drink equivalent chart and will answer questions about their typical alcohol consumption quantity (in standard drink units) on weekdays and weekend days, typical drinking frequency (number of consumption days per week) on weekdays and weekend days, and the highest number of standard drinks consumed at a single occasion during the prior 3 months. If participants work unusual schedules, they will be asked to define the weekend as their day or days off from work. If participants report periods of abstinence and periods of drinking in the previous 3 months, the questions will pertain to periods of drinking. Scores will not be reported on a scale, so there are no minimum and maximum values to report.

SECONDARY OUTCOMES:
Revised Conflict Tactics Scales (CTS2) | Baseline, post-treatment, three-month, six-month, nine-month, and twelve-month follow-ups
  Intimate partner violence (IPV) will be measured using the CTS2, administered to the client regarding their IPV at baseline and follow-up assessments. We will administer only the Physical Assault (12 items) and Psychological Aggression (8 items) subscales to limit respondent burden and because these are most relevant to study hypotheses. The minimum value is 0 and the maximum value is 8. Higher scores represent higher rates of IPV, except for 7 and 8, which represent year and lifetime use and experience of IPV. Variety scores will be calculated for the CTS2 so that scores reflect the number of positively endorsed IPV behaviors (rather than estimates of IPV frequency). This scoring method is considered more reliable, less skewed, more balanced (since high frequency, less severe aggressive behaviors may outweigh the influence of more severe but less frequent violence), and less influenced by recall errors than other methods.

CONTACTS AND LOCATIONS:
Overall Officials: Casey Tyler Taft, PhD, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (3):
- United States (3):
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Strength at Home website — http://www.strengthathome.org